CLINICAL TRIAL: NCT06879561
Title: Impact of Pressure Wire-guidance Versus Angiography-guidance for Infrapopliteal Artery Interventions on Post-procedural Perfusion Status and Wound Healing in Patients With Chronic Limb Threatening Ischemia (PERFECT-CLI)
Brief Title: Pressure Wire Guidance for Infrapopliteal Artery Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2024-0068
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography-guided angioplasty (Active Comparator): In this group, balloon angioplasty will be performed on the target infrapopliteal artery lesion to achieve an optimal procedural result, as determined by angiography. Optimal results are defined as antegrade blood flow without residual stenosis >50% or any flow-limiting dissection.
  Interventions: Procedure: Angiography-guided angioplasty
- Pressure wire-guided angioplasty (Experimental): In this gorup, balloon angioplasty will be performed on the target infrapopliteal artery lesions to achieve an optimal procedural result, as determined by the pressure gradient across the target lesion. An optimal procedural result is defined as pressure gradient less than 10 mmHg, measured using a Pressure Wire.
  Interventions: Procedure: Pressure wire-guided angioplasty

INTERVENTIONS:
Procedure: Angiography-guided angioplasty — Balloon angioplasty will be performed on the target infrapopliteal artery lesion to achieve an optimal procedural result, as determined by angiography. Optimal results are defined as antegrade blood flow without residual stenosis >50% or any flow-limiting dissection.
  Arms: Angiography-guided angioplasty
Procedure: Pressure wire-guided angioplasty — Balloon angioplasty will be performed on the target infrapopliteal artery lesions to achieve an optimal procedural result, as determined by the pressure gradient across the target lesion. An optimal procedural result is defined as pressure gradient less than 10 mmHg, measured using a Pressure Wire.
  Arms: Pressure wire-guided angioplasty

SUMMARY:
"• A prospective, single-center randomized controlled comparison trial.

* A total of 100 patients with symptoms of chronic limb-threatening ischemia (Rutherford category 5) undergoing endovascular treatment for anterior tibial artery or posterior tibial artery lesions will be included if they meet the inclusion criteria and do not meet any exclusion criteria.
* Patients will be randomized in a 1:1 open-label manner either to the pressure wire-guided group or the angiography-guided group.
* Patients will be treated with balloon angioplasty for anetrior tibial artery or posterior tibial artery lesions.
* In the angiography-guided group, balloon angioplasty will be performed to achieve an optimal procedural result, as determined by angiography. Optimal results are defined as antegrade blood flow without residual stenosis >50% or flow-limiting dissection.
* In the Pressure Wire-guided gorup, balloon angioplasty will be performed to obtain optimal procedural result based on both angiography and a pressure gradient over the target lesion. Optimal pressure gradient is less than 10 mmHg by measurement using a Pressure Wire.
* The primary efficacy endpoint is defined by attaiment of skin perfusion pressure ≥50 mmHg within 1-3 days after the index procedure.
* Patients will be followed at 1, 3, and 6 months after the procdure to assess wound healing status, and clinical events."

DETAILED DESCRIPTION:
1. Prospective, singlecenter, open label, randomized controlled study
2. Eligible patients with chronic limb-threatening ischemia (Rutherford category 5) undergoing endovascular treatment for anterior tibial artery or posterior tibial artery lesions will be randomized to pressure wire-guided or angiography-guided groups.
3. All patients will undergo balloon angioplasty for anterior or posterior tibial artery lesions, with the angiography-guided group aiming for optimal procedural results based on angiography, and the pressure wire-guided group aiming for optimal results based on both angiography and pressure gradient measurements.
4. The primary efficacy endpoint is attainment of skin perfusion pressure ≥50 mmHg within 1-3 days after the procedure.
5. Clinical follow-up will occur at 1, 3, and 6 months to assess wound healing and clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic limb threatening ischemia (Rutherford 5)
* Anterior tibial artery or posterior tibial artery lesions ≥ 10 cm Age ≥19 years

Exclusion Criteria:

* Acute limb ischemia
* Contraindication to antiplatelet or anticoagulation agents:

  1. Thrombocytopenia (platelet <100,000/uL)
  2. Previous cerebral hemorrhage, GI bleeding, other reasons for increased bleeding risk within 6 months
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-12-29 (Estimated); Study Completion 2028-08-29 (Estimated)

PRIMARY OUTCOMES:
Attainment rate of postprocedural skin perfusion pressure ≥50 mmHg | Attainment rate of postprocedural skin perfusion pressure≥50 mmHg within 3 days after the indez endovascular therapy
  within 3 days after the index endovascular therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular hospital Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No